CLINICAL TRIAL: NCT03186521
Title: Impact of a Nurse Implemented Sedation and Analgesia Algorithm on Complications of Critical Illness and Outcome of Surgical Intensive Care Patients
Brief Title: Impact of a Nurse Implemented Sedation and Analgesia Algorithm in Surgical Intensive Care Unit
Acronym: ALGOSEDA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 15-147
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Sedation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To show that the nurse implementation of a sedation and analgesia algorithm is beneficial to the patient in terms of sedative drugs reduction and thus overall decrease in duration of mechanical ventilation and the morbidity and mortality which is associated with it, without altering patient comfort and tolerance of the environment. This, compared to the less frequent assessments by doctors and thus regular adjustments during the day as opposed to a fixed drug dose.

DETAILED DESCRIPTION:
Outcome Measures : The primary objective of this non-invasive, non-interventional study is to show that the establishment of a titration algorithm for sedation and analgesia administered by nurses is more beneficial to the patient than the use of such a drug without a suitable regimen. The goal is to improve the quality of our painkillers and sedative drugs use needed in the intensive care environment in order to decrease the morbidity and mortality associated with it, without altering patient comfort and tolerance to the environment. For this we propose to collect a database including patient demographic details, pharmacological information and any possible complications during the ICU stay as well as a distant assessment exploring the psychological complications (3, 6 months and 1 year). The primary endpoint will be the duration of mechanical ventilation, and secondary endpoints, the length of stay in ICU and in hospital, mortality and other complications.

Methods: The two study populations will be in two distinct time periods, the first so-called control without any modification of practices, and the second, by introducing the algorithm with the same drugs being used. Quantitative comparisons of data following a normal distribution will be done using a Student's t test. Otherwise quantitative data will be compared using a Mann-Whitney test or Wilcoxon. The comparison of qualitative data will be done using a Fisher exact test. To increase the power of this before / after study, we calculated the number of patients to be included by period, based on the reduction in duration of mechanical ventilation with such protocols in the literature, and the mean duration of mechanical ventilation in our unit before the study.

ELIGIBILITY:
Inclusion Criteria:

* Any patient sedated, intubated, ventilated whose anticipated duration of sedation is more than 48 hours.
* Age greater than 18 years.

Exclusion Criteria:

* Patient under guardianship or <18.
* Comatose, intracranial hypertension, brain damage, Acute respiratory distress syndrom, acute severe asthma (therapeutic sedation), Post Cardiac Arrest care, Pregnancy
* Neuromuscular blocking agents at the time of inclusion

Secondary Exclusion criteria:

* Extubation <48 hours after inclusion
* Deaths <48 hours after inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients under sedation predicted to last 48hrs or more and aged over 18 years can be included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | baseline
  Duration between endotracheale intubation and extubation

CONTACTS AND LOCATIONS:
Overall Officials: Véronique POTTIER, MD, Principal Investigator — department of anesthesia and intensive care, caen university hospital
Locations (1):
- POTTIER, Caen, France

IPD SHARING:
Plan to Share IPD: No